CLINICAL TRIAL: NCT03899688
Title: Cone Beam Computed Tomography and Histomorphometric Assessments on the Influence a Collagen Membrane Placed on the Antrostomy After Maxillary Sinus Floor Augmentation. A Randomized Clinical Trial.
Brief Title: Tomographic and Histologic Assessment on the Influence of the Use of a Collagen Membrane to Protect the Antrostomy After Maxillary Sinus Floor Augmentation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARDEC Academy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBCT
Record Dates: First submitted 2019-03-23; First posted 2019-04-02 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Alveolar Bone Loss; Alveolar Bone Resorption
Keywords: antrostomy; Maxillary sinus augmentation; collagen membrane; biomaterial
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: test and control group
Who Masked: Investigator, Outcomes Assessor
Masking Description: the surgeon will be blinded until the maxillary sinus augmentation is filled with the biomaterial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test site (Experimental): The space obtained underneath the sinus mucosa will be filled with the xenograft without protecting the antrostomy with a collagen membrane in the test sites. Bone to implant contact was measured at the turned and machined surface.
  Interventions: Procedure: Maxillary sinus augmentation
- control site (Active Comparator): The space obtained underneath the sinus mucosa will be filled with the xenograft and a resorbable collagen membrane will be placed to cover the antrostomy only at the randomly selected control sites. Bone to implant contact was measured at the turned and machined surface.
  Interventions: Procedure: Maxillary sinus augmentation

INTERVENTIONS:
Procedure: Maxillary sinus augmentation — Surgical technique for increasing the vertical bone height of the posterior maxilla an antrostomy of about 5 mm in height and 10 mm long will be prepared using a diamond insert mounted on a sonic-air surgical instrument. The Schneiderian membrane will be elevated and clinical measurements will be performed using an UNC 15 probe. The space obtained underneath the sinus mucosa will be filled with the xenograft and a resorbable collagen membrane will be placed to cover the antrostomy only at the randomly selected control sites.
  Other Names: maxillary sinus lift, maxillary sinus elevation

SUMMARY:
the aim of the present study was to evaluate the dimensional variation and osseointegration of mini-implants at augmented sinus with the antrostomy left unprotected or protected with a collagen membrane.

DETAILED DESCRIPTION:
The Schneiderian mucosa will be elevated and the created space will be filled with a natural bovine bone grafting material (Cerabone® 1-2 mm, Botiss Biomaterials GmbH). In ten patients randomly selected (control sties), a native collagen membrane made of porcine dermis (Collprotect®, Botiss Biomaterials GmbH) will be placed on the antrostomy. In another ten patients of the test group, the antrostomy will be left without the membrane. The flaps will be sutured and anti-inflammatory drugs and antibiotics will be administrated to the patients. The sutures will be removed after 7 days. After 6 months of healing, two mini-implants with different surface will be installed and retrieved after further 3 months for histomorphometric evaluations.

CBCTs will be taken for all patients before surgery (T0), after 1 week from sinus floor augmentation (T1) and after 9 months of healing (T2) and evaluation of dimensional variations over time of soft and hard tissues will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an edentulous atrophic zone in the posterior segment of the maxilla
* Height of the sinus floor ≤4 mm.
* Desiring a prosthetic restoration of the zone using a fix prosthesis supported by implants
* ≥ 21 years of age
* Good general health
* No contraindication for oral surgical procedures
* Not being pregnant.

Exclusion Criteria:The patients will be excluded if they present:

* A systemic disordered.
* Had a chemotherapic or radiotherapeutic treatment.
* Are smokers >10 cigarettes per day
* Have an acute or a chronic sinusitis.
* Had a previous bone augmentation procedures in the zone of interest.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity
Enrollment: 20 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Changing in height of the elevated zone. | The CBCTs will be taken before surgery (T0) and 1-week (T1) and 9 months (T2) after surgery
  will be assessed in the medial, middle and lateral regions of the elevated zone using the cone beam computerized tomographies
Bone-to-implant contact between the different surfaces and between membrane / no membrane groups | three months of healing
  Measurements of new bone formation will be assessed on the histological images taken from the slides and performed between the most coronal bone contact to the surface and the apex of the mini-implant. Comparisons among test and control (without or with a collagen membrane of the access window) and between the two different surface conformations will be performed

SECONDARY OUTCOMES:
Changing in area of the elevated zone | The CBCTs will be taken before surgery (T0) and 1-week (T1) and 9 months (T2) after surgery
  The area will be delineated by the sinus bone walls and the sinus mucosa. The changes will be evaluated on the cone beam computerized tomographies (CBCTs) taken in various periods.
Bone density | three months of healing
  Measurements of new bone formation will be assessed on the histological images taken from the slides and performed between the most coronal bone contact to the surface and the apex of the mini-implant. Comparisons among test and control (without or with a collagen membrane of the access window) and between the two different surface conformations will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Colombia, Cartagena, Cartagena, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852
- [Result] Barone A, Ricci M, Grassi RF, Nannmark U, Quaranta A, Covani U. A 6-month histological analysis on maxillary sinus augmentation with and without use of collagen membranes over the osteotomy window: randomized clinical trial. Clin Oral Implants Res. 2013 Jan;24(1):1-6. doi: 10.1111/j.1600-0501.2011.02340.x. Epub 2011 Dec 12. PMID 22151577
- [Result] Masuda K, Silva ER, Botticelli D, Apaza Alccayhuaman KA, Xavier SP. Antrostomy Preparation for Maxillary Sinus Floor Augmentation Using Drills or a Sonic Instrument: A Microcomputed Tomography and Histomorphometric Study in Rabbits. Int J Oral Maxillofac Implants. 2019 July/August;34(4):819-827. doi: 10.11607/jomi.7350. Epub 2019 Feb 15. PMID 30768660
- [Result] Lundgren S, Andersson S, Gualini F, Sennerby L. Bone reformation with sinus membrane elevation: a new surgical technique for maxillary sinus floor augmentation. Clin Implant Dent Relat Res. 2004;6(3):165-73. PMID 15726851
- [Result] Cricchio G, Sennerby L, Lundgren S. Sinus bone formation and implant survival after sinus membrane elevation and implant placement: a 1- to 6-year follow-up study. Clin Oral Implants Res. 2011 Oct;22(10):1200-1212. doi: 10.1111/j.1600-0501.2010.02096.x. PMID 21906186
- [Result] Moon YS, Sohn DS, Moon JW, Lee JH, Park IS, Lee JK. Comparative histomorphometric analysis of maxillary sinus augmentation with absorbable collagen membrane and osteoinductive replaceable bony window in rabbits. Implant Dent. 2014 Feb;23(1):29-36. doi: 10.1097/ID.0000000000000031. PMID 24445918
- [Result] Omori Y, Ricardo Silva E, Botticelli D, Apaza Alccayhuaman KA, Lang NP, Xavier SP. Reposition of the bone plate over the antrostomy in maxillary sinus augmentation: A histomorphometric study in rabbits. Clin Oral Implants Res. 2018 Aug;29(8):821-834. doi: 10.1111/clr.13292. Epub 2018 Jun 7. PMID 29876969
- [Result] Corbella S, Taschieri S, Weinstein R, Del Fabbro M. Histomorphometric outcomes after lateral sinus floor elevation procedure: a systematic review of the literature and meta-analysis. Clin Oral Implants Res. 2016 Sep;27(9):1106-22. doi: 10.1111/clr.12702. Epub 2015 Oct 10. PMID 26452326
- [Result] Caneva M, Lang NP, Garcia Rangel IJ, Ferreira S, Caneva M, De Santis E, Botticelli D. Sinus mucosa elevation using Bio-Oss(R) or Gingistat(R) collagen sponge: an experimental study in rabbits. Clin Oral Implants Res. 2017 Jul;28(7):e21-e30. doi: 10.1111/clr.12850. Epub 2016 Apr 15. PMID 27080163
- [Result] De Santis E, Lang NP, Ferreira S, Rangel Garcia I Jr, Caneva M, Botticelli D. Healing at implants installed concurrently to maxillary sinus floor elevation with Bio-Oss(R) or autologous bone grafts. A histo-morphometric study in rabbits. Clin Oral Implants Res. 2017 May;28(5):503-511. doi: 10.1111/clr.12825. Epub 2016 Mar 10. PMID 26969193
- [Result] Riachi F, Naaman N, Tabarani C, Aboelsaad N, Aboushelib MN, Berberi A, Salameh Z. Influence of material properties on rate of resorption of two bone graft materials after sinus lift using radiographic assessment. Int J Dent. 2012;2012:737262. doi: 10.1155/2012/737262. Epub 2012 Jul 31. PMID 22899930
- [Result] Shanbhag S, Shanbhag V, Stavropoulos A. Volume changes of maxillary sinus augmentations over time: a systematic review. Int J Oral Maxillofac Implants. 2014 Jul-Aug;29(4):881-92. doi: 10.11607/jomi.3472. PMID 25032768

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT03899688/Prot_SAP_001.pdf